CLINICAL TRIAL: NCT00029497
Title: Sham Device, Pill Placebo or Treatment For Arm Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: R01AT000402-01 (NIH)
Record Dates: First submitted 2002-01-14; First posted 2002-01-15 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Cumulative Trauma Disorders; Repetitive Strain Injury; Carpal Tunnel Syndrome; Pain
MeSH Terms: conditions — Cumulative Trauma Disorders; Carpal Tunnel Syndrome; Pain | interventions — Acupuncture Therapy; Amitriptyline

INTERVENTIONS:
Procedure: Acupuncture
Drug: Amitriptyline

SUMMARY:
This study investigates the role of two active interventions and their placebo effects in randomized control trials. The study conducts two parallel trials of treatments for upper extremity pain secondary to repetitive stress disorder, including carpal tunnel syndrome. The active interventions are amitriptyline and acupuncture. The placebo are sham acupuncture device and placebo pill.

DETAILED DESCRIPTION:
There is evidence that the magnitude of the placebo effect produced by a device is greater than that produced by a pill. If this is the case, it has significant ramifications for all trials involving devices and for our understanding of the role of the placebo effect in randomized controlled trials (RCT). This two phase study 1)investigates the role of the placebo effect in RCT's and 2)conducts two trials of treatments for persistent upper extremity pain secondary to repetitive strain injury (RSI), including carpel tunnel syndrome. In Phase I. 240 patients with RSI are randomly assigned to receive a placebo device (a recently validated sham acupuncture device) or a placebo pill (dummy amitriptyline). Our primary hypothesis is that patients will respond better to the sham device than the placebo pill. A finding that sham acupuncture produces a greater placebo response than a placebo pill has important implications for the interpretation of results in trials that compare devices to sham devices, devices to pills, and medical management to surgery. Phase II randomly assigns patients from the sham acupuncture arm of Phase I to receive either TCA or continue to receive the sham version. Patients in the placebo pill arm of Phase I will be randomly assigned to receive either AMI or continue receiving the placebo pill. From the patients'perspective, the shift in treatment assignment from Phase I to II should not be noticeable. Phase II will allow us to test whether the active treatments outperform their respective placebos. Both of these treatments have shown promise in small studies, but neither has been prospectively studied in a large trial with appropriate controls. Because Phase I also functions as a run-in period for Phase II, analysis combining both phases will allow us to examine whether a run-in has methodological advantages in a device trial. Moreover, combined analyses permit testing whether patients level of response to placebo in Phase I affects their response to active treatment Phase II. A positive finding here would contribute importantly to our understanding of the role of the placebo in RCTs.

ELIGIBILITY:
Inclusion Criteria:

* Treated for repetitive strain injury for at least 3 months at a clinical site in the Greater Boston Area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ted Kaptchuk, OMD, Principal Investigator — Harvard
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cambridge Hospital, Cambridge, Massachusetts